CLINICAL TRIAL: NCT01230931
Title: Hemostasis in Kocher-Langenbeck Approaches for Acetabular Surgery Using a Topical Surgical Hemostat
Brief Title: Hemostasis in Kocher-Langenbeck Approaches for Acetabular Surgery Using a Topical Surgical Hemostat (Vitagel)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team left institution; no one remaining to finish study
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Catherine G. Ambrose, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-09-0654
Record Dates: First submitted 2010-10-18; First posted 2010-10-29 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Fracture Fixation; Intra-Articular Fractures; Acetabulum
Keywords: Acetabulum; Fracture; Hemostatis; Vitagel; Fibrin sealant
MeSH Terms: conditions — Intra-Articular Fractures; Fractures, Bone | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vitagel and Standard of Care (Experimental): This group of patients will receive the vitagel topical surgical hemostat spray intra-operatively, along with all the other standards of care.
  Interventions: Device: Vitagel; Procedure: Standard of care
- Standard of Care (Active Comparator): This group of patients will receive the standard of care for hemostasis in acetabular surgery (electrocautery/ligation of bleeding vessels, fracture reduction and stabilization, cell-saver, lap packing). They will not receive the vitagel product.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: Vitagel — Vitagel (by Stryker) is a topical surgical hemostat spray that results in coagulation. The components are as follows: autogenous blood is drawn and centrifuged to produce a sample of platelets and growth factors; this is combined with a bovine thrombin and collagen solution. When the two are applied together, it produces the hemostatic effect.
  Arms: Vitagel and Standard of Care
Procedure: Standard of care — Standard of care for hemostasis in acetabular surgery includes electrocautery/ligation of bleeding vessels, fracture reduction and stabilization, cell-saver, lap packing.

SUMMARY:
The purpose of the study is to determine whether surgical hemostats can minimize blood loss, need for allogeneic blood transfusions and their associated risks, and costs in patients with certain acetabular fractures requiring operative fixation via a non-extensile Kocher-Langenbeck surgical approach. Since surgical hemostats and other topical agents like platelet gel products have also been linked with improved wound healing, incidence of wound dehiscence and/or infections will also be examined. The investigators primary hypothesis is the topical hemostat will result in lower blood losses intraoperatively and fewer units of perioperative blood product transfused.

ELIGIBILITY:
Inclusion Criteria:

* Acetabular fracture deemed to require open reduction and internal fixation by one of the three principle attending surgeons.
* Fixation must require a single non-extensile posterior approach (Kocher-Langenbeck)
* Posterior wall, Posterior column, certain simple transverse and transverse associated with a posterior wall, T-type, and posterior wall-posterior column fracture types
* Ages 18-65
* Patient or family must consent to the research protocol

Exclusion Criteria:

* Not meeting the aforementioned inclusion criteria
* Unstable hemoglobin levels for three days prior to acetabular surgery (i.e. no other bleeding sources)
* Revision surgery
* Surgery occurring more than two weeks post-injury
* History of blood dyscrasias or immunocompromised patients
* Patients with medical conditions requiring anticoagulation or international normalized ratio (INR) above 1.5
* Obese patients (BMI >35)
* Known ongoing infection (local or systemic)
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine G Ambrose, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Thoms RJ, Marwin SE. The role of fibrin sealants in orthopaedic surgery. J Am Acad Orthop Surg. 2009 Dec;17(12):727-36. doi: 10.5435/00124635-200912000-00001. PMID 19948697
- [Background] Gardner MJ, Demetrakopoulos D, Klepchick PR, Mooar PA. The efficacy of autologous platelet gel in pain control and blood loss in total knee arthroplasty. An analysis of the haemoglobin, narcotic requirement and range of motion. Int Orthop. 2007 Jun;31(3):309-13. doi: 10.1007/s00264-006-0174-z. Epub 2006 Jul 1. PMID 16816947
- [Background] Zavadil DP, Satterlee CC, Costigan JM, Holt DW, Shostrom VK. Autologous platelet gel and platelet-poor plasma reduce pain with total shoulder arthroplasty. J Extra Corpor Technol. 2007 Sep;39(3):177-82. PMID 17972452
- [Background] Everts PA, Devilee RJ, Brown Mahoney C, Eeftinck-Schattenkerk M, Box HA, Knape JT, van Zundert A. Platelet gel and fibrin sealant reduce allogeneic blood transfusions in total knee arthroplasty. Acta Anaesthesiol Scand. 2006 May;50(5):593-9. doi: 10.1111/j.1399-6576.2006.001005.x. PMID 16643230
- [Background] Horstmann WG, Slappendel R, van Hellemondt GG, Wymenga AW, Jack N, Everts PA. Autologous platelet gel in total knee arthroplasty: a prospective randomized study. Knee Surg Sports Traumatol Arthrosc. 2011 Jan;19(1):115-21. doi: 10.1007/s00167-010-1207-0. Epub 2010 Jul 18. PMID 20640848
- [Background] Wang GJ, Hungerford DS, Savory CG, Rosenberg AG, Mont MA, Burks SG, Mayers SL, Spotnitz WD. Use of fibrin sealant to reduce bloody drainage and hemoglobin loss after total knee arthroplasty: a brief note on a randomized prospective trial. J Bone Joint Surg Am. 2001 Oct;83(10):1503-5. doi: 10.2106/00004623-200110000-00007. PMID 11679600
- [Background] Wang GJ, Goldthwaite CA Jr, Burks S, Crawford R, Spotnitz WD; Orthopaedic Investigators Group. Fibrin sealant reduces perioperative blood loss in total hip replacement. J Long Term Eff Med Implants. 2003;13(5):399-411. doi: 10.1615/jlongtermeffmedimplants.v13.i5.50. PMID 14649578
- [Background] Sherman R, Chapman WC, Hannon G, Block JE. Control of bone bleeding at the sternum and iliac crest donor sites using a collagen-based composite combined with autologous plasma: results of a randomized controlled trial. Orthopedics. 2001 Feb;24(2):137-41. doi: 10.3928/0147-7447-20010201-16. PMID 11284596
- [Background] Levy O, Martinowitz U, Oran A, Tauber C, Horoszowski H. The use of fibrin tissue adhesive to reduce blood loss and the need for blood transfusion after total knee arthroplasty. A prospective, randomized, multicenter study. J Bone Joint Surg Am. 1999 Nov;81(11):1580-8. doi: 10.2106/00004623-199911000-00010. PMID 10565650
- [Background] Cillo JE Jr, Marx RE, Stevens MR. Evaluation of autologous platelet-poor plasma gel as a hemostatic adjunct after posterior iliac crest bone harvest. J Oral Maxillofac Surg. 2007 Sep;65(9):1734-8. doi: 10.1016/j.joms.2006.09.008. PMID 17719390
- [Background] Goodnough LT, Brecher ME, Kanter MH, AuBuchon JP. Transfusion medicine. First of two parts--blood transfusion. N Engl J Med. 1999 Feb 11;340(6):438-47. doi: 10.1056/NEJM199902113400606. No abstract available. PMID 9971869
- [Background] Busch MP, Kleinman SH, Nemo GJ. Current and emerging infectious risks of blood transfusions. JAMA. 2003 Feb 26;289(8):959-62. doi: 10.1001/jama.289.8.959. No abstract available. PMID 12597733
- See also: UT-Houston Department of Orthopaedic Surgery — https://med.uth.edu/ortho/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 were enrolled, but only 20 were randomized.
Groups:
- Vitagel and Standard of Care: The group of patients will receive the vitagel topical surgical hemostat spray intra-operatively, along with all the other standards of care.
  Vitagel: Vitagel (by Stryker) is a topical surgical hemostat spray that results in coagulation. The components are as follows: autogenous blood is drawn and centrifuged to produce a sample of platelets and growth factors; this is combined with a bovine thrombin and collagen solution. When the two are applied together, it produces the hemostatic effect.
  Standard of care: Standard of care for hemostasis in acetabular surgery includes electrocautery/ligation of bleeding vessels, fracture reduction and stabilization, cell-saver, lap packing.
Period: Overall Study
Arm/Group | Vitagel and Standard of Care | Standard of Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitagel and Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.7) | 36.4 (8.5) | 33.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Rate of Blood Volume Loss
Description: The amount of blood loss during the surgery as measured by cell saver and lap counts. The cell saver and lap count totals will be summed.
Time Frame: at the time of surgery
Measure: Mean (Standard Deviation); unit: milliliters per minute (mL/min)
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
milliliters per minute (mL/min) | 2.65 (1.43) | 3.63 (3.85)

2. Secondary Outcome: Change in Hemoglobin Level
Description: The amount of change in hemoglobin level from before surgery on the operative day until post-operative day numbers one, two, or three.
Time Frame: baseline, post-operative day 1
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
grams per deciliter (g/dL) | -1.05 (1.25) | -1.16 (1.46)

3. Secondary Outcome: Change in Hemoglobin Level
Description: as for outcome 2
Time Frame: baseline, post-operative day 2
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
grams per deciliter (g/dL) | -1.23 (1.33) | -1.41 (1.72)

4. Secondary Outcome: Change in Hemoglobin Level
Description: as for outcome 2
Time Frame: baseline, post-operative day 3
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
grams per deciliter (g/dL) | -1.12 (1.60) | -1.52 (1.86)

5. Secondary Outcome: Volume of Blood Products Transfused
Description: The amount of blood products [packed red blood cells (pRBCs), fresh frozen plasma (FFP), intra-operative salvaged blood collected with a cell saver] transfused will be recorded throughout the operative day and on post-operative days 1, 2, and 3.
Time Frame: baseline through post-operative day 3
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
milliliters | 455 (554) | 675 (1362)

6. Secondary Outcome: Units of Packed Red Blood Cells (pRBCs) Transfused
Description: as for outcome 5
Time Frame: baseline through post-operative day 3
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
units | 0.8 (1.3) | 1.0 (2.2)

7. Secondary Outcome: Units of Fresh Frozen Plasma (FFP) Transfused
Description: The amount of blood products (pRBCs and FFP) transfused will be recorded throughout the operative day and on post-operative days 1, 2, and 3. Intra-operative salvaged blood will be recovered with a cell saver, and if cell saver units are transfused, this will also be recorded on the operative day and on post-operative days 1, 2, and 3.
Time Frame: baseline through post-operative day 3
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
units | 0.10 (0.32) | 0.40 (0.97)

8. Secondary Outcome: Volume of Intra-operative Salvaged Blood Transfused
Description: as for outcome 7
Time Frame: baseline through post-operative day 3
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
milliliters | 175 (168.7) | 325 (697.7)

9. Secondary Outcome: Number of Participants With a Wound Complication
Description: The number of wound complications (dehiscence, infection) or the need to return to the operating to address a wound complication will be recorded. Wound complications will be recorded from the day of surgery until an average of two weeks post-operatively (this study is an acute care study, so no data will be collected after the initial hospital stay).
Time Frame: at the time of discharge (about 2 weeks after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Vitagel and Standard of Care | Standard of Care
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Through the hospital stay (average length of stay was 11.5 days, range was 5-24 days)
Description: The below-listed Adverse Events were not related to the intervention under study.
Arm/Group | Vitagel and Standard of Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitagel and Standard of Care (N=10) | Standard of Care (N=10)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Deep Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Ischemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes